CLINICAL TRIAL: NCT05923528
Title: Comparison of Non-pharmaceutical Treatments for Evaporative Dry Eye: A Randomized Controlled Study
Brief Title: Comparison of Non-pharmaceutical Treatments for Evaporative Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TREATDE2023
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-06

CONDITIONS: Dry Eye
Keywords: dry eye; intense pulsed light; heated eye mask; eyepeace; lipiflow
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: IPL group (Experimental): participants will receive IPL treatment with 12 homogeneously spaced pulses of light to both eyes at day 0, day 14, and day 28
  Interventions: Device: IPL
- Group B: HEM group (Experimental): participants were applied an air-activated disposable eye mask on both closed eyes (Ocuface Medical Co., Ltd., Guangzhou, China) simultaneously for 15 minutes according to the manufacturer's instructions every day for 42 days
  Interventions: Device: Heated eye mask
- Group C: VTPS group (Experimental): VTPS group, Patients will receive a single 12-minute treatment using the LipiFlow® (TearScience Inc., Morrisville, NC) on both eyes at day 0
  Interventions: Device: LipiFlow®
- Group D: EyePeace® group (Experimental): Participants were followed immediately by 10 gentle squeezes of the eyelid massage device (EMD) on both eyes, and 10 gentle eyelid massaging movements using the index and middle fingers every day for 42 days.
  Interventions: Device: EyePeace®

INTERVENTIONS:
Device: IPL — IPL treatment intensity was chosen based on the Fitzpatrick scale as follows: Fitzpatrick scale I, II, III, 10-15 J/cm2 with a 570-nm filter
  Arms: Group A: IPL group
Device: Heated eye mask — Heated eye mask will be used to assess its usefulness in dry eye signs and symptoms
  Arms: Group B: HEM group
Device: LipiFlow® — LipiFlow® can control the variables of temperature, pressure, and MG expression technique
  Arms: Group C: VTPS group
Device: EyePeace® — The silicone-made flexible hand-held gadget applies regulated, vertical pressure to the closed eyelids.
  Arms: Group D: EyePeace® group

SUMMARY:
The lipid layer of the tear film is critical to maintaining the integrity of the tear film and deficiency in the tear film lipid layer (TFLL) is the cause of evaporative dry eye (EDE) in approximately 80% of dry eye disease patients, resulting in excessive evaporation (so-called hyperevaporative dry eye). This study protocol was designed to assess and compare the effects of intense pulsed light (IPL), heated eye mask (HEM), vectored thermal pulsation system (VTPS), and eyelid massage device (EMD) for improving signs and symptoms of EDE.

EDE patients will be randomly divided into IPL, HEM, VTPS, and EMD groups and will be followed up for four weeks. The primary outcome measure will be non-invasive tear breakup time (NITBUT). The secondary outcome measures will include, tear film lipid layer score (TFLL), meibomian gland function and secretion quality change from baseline conjunctival and cornea staining (CFS) with fluorescein and lissamine, tear meniscus height (TMH), conjunctival hyperemia (RS score) and ocular surface disease index (OSDI) questionnaire. Additionally, adverse events also were monitored and documented.

DETAILED DESCRIPTION:
"A chronic, diffuse abnormality of the meibomian glands, frequently characterized by terminal duct obstruction and/or qualitative/quantitative abnormalities in glandular secretion," is how the International Workshop on meibomian gland (MG) hypofunction or dysfunction (MGD) describes MGD. These glands, which are repurposed sebaceous glands, secrete meibum onto the ocular surface. By improving the quality and quantity of meibum secretion, signs and symptoms of evaporative dry eye (EDE) and MGD can be alleviated.

Traditional remedies derived from natural sources have been utilized for treating anterior eye ailments since ancient times, predating the advent of contemporary pharmacological interventions. These remedies continue to be employed in diverse populations globally. The objective of this study is to examine the present non-pharmacological modalities that have been implemented and evaluate their efficacy. This encompasses alternative medicine, extant non-pharmaceutical therapeutic modalities, as well as contemporary low and high technological interventions. The most common approaches to relieving MGD involve the application of heat to the eyelids with and without physical massage of the eyelids in order to express the MGs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able and willing to comply with the treatment/follow-up schedule
* Bilateral signs and symptoms of dry eye disease (a) the ocular surface disease index (OSDI) questionnaire ≥ 13, (b) a non-invasive tear film breakup time (NITBUT) of ≤10 s, or a conjunctivocorneal staining score (CS) of ≥ 3 points. The presence of two or more criteria was used to establish a positive DE diagnosis, based on the 2016 Asia Dry Eye Society criteria
* Lipid layer thickness score evaluation ≥ 2.

Exclusion Criteria:

* existing ocular trauma, infectious diseases, recent surgical history
* skin defects, pigmentation, moles, scars in the treatment area, skin cancer
* autoimmune diseases, skin allergies
* pregnancy or lactation
* photophobia that may cause reflex tearing or difficulty in evaluating the patient's lipid layer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-invasive tear breakup time (NITBUT) | • Changes at day-14, day-28 and day-42will be compare with baseline measurements. • Comparison between groups at baseline, day-14, day-28 and day-42will also be examined.
  Non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequential readings will be captured, and the median value will be included in the final analysis. The median value will be recorded

SECONDARY OUTCOMES:
Tear Film Lipid Layer Score (TFLL) | • Changes at day-14, day-28 and day-42will be compare with baseline measurements. • Comparison between groups at baseline, day-14, day-28 and day-42will also be examined.
  Tear film lipid layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan). The results will be graded as follows: grade 1, somewhat gray color, uniform distribution; grade 2, somewhat gray color, nonuniform distribution; grade 3, a few colors, nonuniform distribution; grade 4, many colors, nonuniform distribution; grade 5, corneal surface partially exposed
Meibomian gland function and secretion quality | • Changes at day-14, day-28 and day-42will be compare with baseline measurements. • Comparison between groups at baseline, day-14, day-28 and day-42will also be examined.
  Five meibomian glands in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste-like consistency meibum)
Ocular Surface Disease Index (OSDI) | • Changes at day-14, day-28 and day-42will be compare with baseline measurements. • Comparison between groups at baseline, day-14, day-28 and day-42will also be examined.
  The patient will answer each question on a scale ranging from 0 to 4, with 0 indicating 'none of the time' and 4 indicating 'all of the time'. If a certain question is deemed irrelevant, it will be marked as 'not applicable (N/A)' and excluded from the analysis. The OSDI total score is calculated according to the following formula. The scale ranges from 0 to 100, with higher scores representing more severe cases of dry eye syndrome
Fluorescein and lissamine conjunctival and cornea staining (CFS) | • Changes at day-14, day-28 and day-42will be compare with baseline measurements. • Comparison between groups at baseline, day-14, day-28 and day-42will also be examined.
  Fluorescein and lissamine staining of the ocular surface will be divided into three zones comprising nasal conjunctival, corneal, and temporal conjunctival areas. The staining score ranged from 0 to 3 for each zone, yielding a total score of 0-9 for the ocular surface
Tear meniscus height (TMH) | • Changes at day-14, day-28 and day-42will be compare with baseline measurements. • Comparison between groups at baseline, day-14, day-28 and day-42will also be examined.
  Non-invasive first tear film breakup time using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively and the median value was recorded
Conjunctival hyperemia (RS score) | • Changes at day-14, day-28 and day-42will be compare with baseline measurements. • Comparison between groups at baseline, day-14, day-28 and day-42will also be examined.
  Conjunctival hyperemia (RS score) will be assessed by Keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 (normal) to 4.0 (severe)
Thermal imaging: Ocular surface temperature (OST) | • Changes at day-14, day-28 and day-42will be compare with baseline measurements. • Comparison between groups at baseline, day-14, day-28 and day-42will also be examined.
  All measurements were taken in the same room with controlled temperature and humidity. Prior to ocular thermography or other tests, participants were acclimatized to the room for 20 minutes. Morgan and colleagues described the following criteria for recording OST: The patients were instructed to blink normally, close their eyes for 3 seconds, and the first image was captured soon after the eyelids opened. The temperature was taken in the central cornea, which was defined as a circular area 4 mm in diameter in the middle of the cornea

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Eric Pazo, Study Chair — He eye specialist hospital

IPD SHARING:
Plan to Share IPD: Yes
The study's findings will be shared regardless of the effect's direction. All possible beneficiaries of the research, including patients, carers, family, doctors, advisory boards, and medical boards, will receive trial data. Publications in high impact, open-access medical journals and talks at national and international medical conferences will serve this purpose.
Supporting Information: Study Protocol, SAP
Time Frame: The Steering Committee will write and submit the report for publication at the end of the study

REFERENCES:
- [Background] Ma J, Pazo EE, Zou Z, Jin F. Prevalence of symptomatic dry eye in breast cancer patients undergoing systemic adjuvant treatment: A cross-sectional study. Breast. 2020 Oct;53:164-171. doi: 10.1016/j.breast.2020.07.009. Epub 2020 Aug 5. PMID 32836200
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Zhang X, Wang L, Zheng Y, Deng L, Huang X. Prevalence of dry eye disease in the elderly: A protocol of systematic review and meta-analysis. Medicine (Baltimore). 2020 Sep 11;99(37):e22234. doi: 10.1097/MD.0000000000022234. PMID 32925801
- [Background] Wu MF, Gao H, Zhao LJ, Chen H, Huang YK. Real dynamic assessment of tear film optical quality for monitoring and early prevention of dry eye. Medicine (Baltimore). 2020 Jul 31;99(31):e21494. doi: 10.1097/MD.0000000000021494. PMID 32756182
- [Background] Fu J, Chou Y, Hao R, Jiang X, Liu Y, Li X. Evaluation of ocular surface impairment in meibomian gland dysfunction of varying severity using a comprehensive grading scale. Medicine (Baltimore). 2019 Aug;98(31):e16547. doi: 10.1097/MD.0000000000016547. PMID 31374018
- [Background] Heidari M, Noorizadeh F, Wu K, Inomata T, Mashaghi A. Dry Eye Disease: Emerging Approaches to Disease Analysis and Therapy. J Clin Med. 2019 Sep 11;8(9):1439. doi: 10.3390/jcm8091439. PMID 31514344
- [Background] Song Y, Yu S, He X, Yang L, Wu Y, Qin G, Zhang Q, Deep Singh Talwar G, Xu L, Moore JE, He W, Pazo EE. Tear film interferometry assessment after intense pulsed light in dry eye disease: A randomized, single masked, sham-controlled study. Cont Lens Anterior Eye. 2022 Aug;45(4):101499. doi: 10.1016/j.clae.2021.101499. Epub 2021 Aug 22. PMID 34433517
- [Background] Ikonne EU, Ikpeazu VO, Ugbogu EA. The potential health benefits of dietary natural plant products in age related eye diseases. Heliyon. 2020 Jul 10;6(7):e04408. doi: 10.1016/j.heliyon.2020.e04408. eCollection 2020 Jul. PMID 32685729
- [Background] Matsumoto Y, Dogru M, Goto E, Ishida R, Kojima T, Onguchi T, Yagi Y, Shimazaki J, Tsubota K. Efficacy of a new warm moist air device on tear functions of patients with simple meibomian gland dysfunction. Cornea. 2006 Jul;25(6):644-50. doi: 10.1097/01.ico.0000208822.70732.25. PMID 17077654
- [Background] Xu L, Wu Y, Song Y, Zhang Q, Qin G, Yang L, Ma J, Palme C, Moore JE, Pazo EE, He W. Comparison Between Heated Eye Mask and Intense Pulsed Light Treatment for Contact Lens-Related Dry Eye. Photobiomodul Photomed Laser Surg. 2022 Mar;40(3):189-197. doi: 10.1089/photob.2021.0094. PMID 35298282
- [Background] Wu Y, Xu L, Song Y, Zhang Q, Qin G, Yang L, Ma J, Palme C, Moore JE, Pazo EE, He W. Management of Post-LASIK Dry Eye with Intense Pulsed Light in Combination with 0.1% Sodium Hyaluronate and Heated Eye Mask. Ophthalmol Ther. 2022 Feb;11(1):161-176. doi: 10.1007/s40123-021-00418-2. Epub 2021 Nov 6. PMID 34741758
- [Background] Olson MC, Korb DR, Greiner JV. Increase in tear film lipid layer thickness following treatment with warm compresses in patients with meibomian gland dysfunction. Eye Contact Lens. 2003 Apr;29(2):96-9. doi: 10.1097/01.ICL.0000060998.20142.8D. PMID 12695712
- [Background] Wang MTM, Feng J, Wong J, Turnbull PR, Craig JP. Randomised trial of the clinical utility of an eyelid massage device for the management of meibomian gland dysfunction. Cont Lens Anterior Eye. 2019 Dec;42(6):620-624. doi: 10.1016/j.clae.2019.07.008. Epub 2019 Jul 26. PMID 31358441
- [Derived] Chen J, Qin G, Yu S, Moore J, Xu L, He W, Pazo EE, He X. Comparison of non-pharmaceutical treatments for evaporative dry eye: a randomised controlled study protocol. BMJ Open. 2024 Feb 26;14(2):e078727. doi: 10.1136/bmjopen-2023-078727. PMID 38413161